CLINICAL TRIAL: NCT04649606
Title: Dynamic Characterisation of Meibomian Gland Structure
Status: Completed | Type: Observational
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CR-6369
Record Dates: First submitted 2020-11-09; First posted 2020-12-02 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2021-07

CONDITIONS: Visual Acuity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Experimental: Eligible subjects will undergo repeated observations to evaluate the Meibomian gland appearance

SUMMARY:
This will be a single center pilot study to evaluate appearance of the Meibomian glands.

ELIGIBILITY:
Inclusion Criteria:

* Potential subjects must satisfy all of the following criteria to be enrolled in the study:

  1. Healthy adult males and females, 18-40 years of age (inclusive)
  2. The subject must read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form
  3. The subject must appear able and willing to adhere to the instructions set forth in this clinical protocol
  4. The subject must agree not to participate in other clinical research for the duration of this study
  5. The subject's optimal spherical equivalent distance refraction must be between +1.00 and -2.00 D in each eye
  6. The subject's refractive cylinder must be ≤-1.00 DC in each eye
  7. The subject must score less than 4 points (inclusive) in SPEED questionnaire

     Exclusion Criteria:
* Potential subjects who meet any of the following criteria will be excluded from participating in the study:

  1. Currently pregnant or lactating
  2. Any systemic disease (e.g. Sjögren's Syndrome), allergies, infectious disease (e.g. hepatitis, tuberculosis), contagious immunosuppressive diseases (e.g. HIV), autoimmune disease (e.g. rheumatoid arthritis), or other diseases, by self-report, which are known to interfere with contact lens wear and/or participation in the study
  3. Have had cataract surgery
  4. Use of systemic medications (e.g. chronic steroid use) and any current use of ocular medications (e.g. lubricants, artificial tears) that would interfere with participation in the trial, at the Investigator's discretion
  5. They have history (more than one week in total) of contact lens wear.
  6. Any previous, or planned (during the course of the study) ocular surgery (e.g. radial keratotomy, PRK, LASIK, etc.)
  7. Any ocular allergies, infections or other ocular abnormalities that are known to interfere with participation in the study. This may include, but not be limited to entropion, ectropion, extrusions, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, aphakia, corneal distortion or keratoconus
  8. History of allergy to sodium fluorescein or lissamine green
  9. Any Grade 1.5 or greater slit lamp findings (e.g. oedema, corneal neovascularization, corneal staining, tarsal abnormalities, conjunctival injection) on the Efron Grading Scales or other ocular abnormality including Meibomian gland dysfunction (MGD) or blepharitis (Grade 1.0 or greater)
  10. Meibomian gland atrophy exceeds 25% (inclusive) in either lower or upper eyelid
  11. The central glands atrophy exceeds 25% (inclusive)
  12. The number of Meibomian glands yielding liquid secretion (MGYLS) is 6 or less (applicable to Phase II subjects only)
  13. Use of eye makeup on the days of the study visits
  14. Participation in any pharmaceutical or medical device related clinical trial within 14 days prior to study enrolment
  15. Employee or immediate family member of an employee of clinical site (e.g. Investigator, Coordinator, Technician)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subjects will be recruited and enrolled based on Inclusion/Exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2020-10-19 (Actual); Primary Completion 2021-06-22 (Actual); Study Completion 2021-06-22 (Actual)

PRIMARY OUTCOMES:
Meibomian Gland Appearance - Area | up to 4-week follow-up
  Meibomian gland appearance will be evaluated on both eyes using a custom image analysis algorithm, which calculates the area corresponding to individual and aggregated Meibomian glands.
Meibomian Gland Appearance - Mean Reflectivity | up to 4-week follow-up
  Meibomian gland appearance will be evaluated on both eyes using a custom image analysis algorithm, which calculates the mean reflectivity of individual and aggregated Meibomian glands

SECONDARY OUTCOMES:
Lipid Layer Thickness (LLT) | up to 4-week follow-up
  LLT will be measured using the LipiView® II instrument on the right eye only.
Non-Invasive Tear Break-Up Time (NIBUT) | up to 4-week follow-up
  NIBUT will be evaluated using the Medmont E300 instrument, with three measurements taken for the right eye only, at least 30 seconds apart and the median recorded.
Tear Film Evaporation Rate | up to 4-week follow-up
  Tear film evaporation rate will be assessed using the Eye-VapoMeter for 3 consecutive open eye measurements followed by 3 consecutive closed eye measurements. The mean for each method will be calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Manchester, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu